CLINICAL TRIAL: NCT00132600
Title: Clinical Evaluation of Bacitracin. A Phase II Dose-Response Study
Brief Title: Clinical Evaluation of Bacitracin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mekos Laboratories AS (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: Mekos 05 P36/2
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2005-10-19 (Estimated); Status verified 2005-08

CONDITIONS: Allergic Contact Dermatitis
Keywords: Allergic contact dermatitis; Patch testing; bacitracin
MeSH Terms: conditions — Dermatitis, Allergic Contact | interventions — Bacitracin; Allergens

INTERVENTIONS:
Drug: bacitracin (allergen)

SUMMARY:
The purpose of this study is to establish a concentration of a bacitracin-patch for diagnosing allergic contact dermatitis.

DETAILED DESCRIPTION:
Thin-layer Rapid Use Epicutaneous Test (T.R.U.E. Test®) is a ready-to-use patch test method designed for diagnosis of allergic contact dermatitis.

The standard panel consists of two tape strips, panel 1, with 11 allergen patches and a negative control and panel 2, with 12 allergen patches. T.R.U.E. TestTM panels 1 and 2 contain 23 of the most frequent contact allergens. With the 23 allergens the test currently consists of, it is possible to detect about 60-70% of contact allergic reactions. Thus, there is a need for expanding the number of allergens included in T.R.U.E.Test in order to detect more contact allergic reactions. Bacitracin is one of these allergens, and the purpose of this study is to determine a concentration for the patch by using a bacitracin dilution series.

ELIGIBILITY:
Inclusion Criteria:

* Positive bacitracin patch test within the latest 5 years.
* Age greater than or equal to 18 years.
* Signed informed consent.

Exclusion Criteria:

* Topical treatment with corticosteroids or immunosuppressives during the latest 7 days on the test area or near the test area.
* Systemic treatment with corticosteroids or immunosuppressives during the latest 7 days.
* Treatment with ultraviolet (UV)-light during the latest 3 weeks.
* Widespread active dermatitis or dermatitis on test area.
* Breast-feeding or pregnancy. Females of childbearing potential must demonstrate a negative pregnancy test before inclusion in the study.
* Subjects not able to cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-04; Study Completion 2005-07

PRIMARY OUTCOMES:
Skin reaction to the patch test after 72-96 hours and after 7 days

SECONDARY OUTCOMES:
Evaluation of safety including late and persistent responses
Evaluation day 3/4, day 7 and day 21

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Fowler, Prof., Principal Investigator — Mekos Laboratories AS
Locations (1):
- Dermatological Clinic (Joseph Fowler MD), Louisville, Kentucky, United States